CLINICAL TRIAL: NCT03206866
Title: Role of Serum Regucalcin in Diagnosis of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed_Elalfy, medical oncology resident, Mansoura University
Other Study IDs: SMP30
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Role of Serum Regucalcin in Diagnosis of HCC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with HCC
  Interventions: Diagnostic Test: serum regucalcin antibody
- patients with hepatitis C Ab positive
  Interventions: Diagnostic Test: serum regucalcin antibody
- patients with hepatitis C Ab negative
  Interventions: Diagnostic Test: serum regucalcin antibody

INTERVENTIONS:
Diagnostic Test: serum regucalcin antibody — serum regucalcin antibody

SUMMARY:
Although the diagnosis and therapy of HCC have being improved, the poor prognosis still remains. To reduce the mortality and improve the effectiveness of diagnosis and therapy, it is important to detect the protein biomarkers which are associated with HCC tumor progression and may be useful as potential diagnosis or therapeutic targets.

SMP30 (senescence marker protein 30)(serum regucalcin), which we have previously identiﬁed from Guangxi HCC cDNA expression library by the SEREX approach, is one of the hepatocellular carcinoma associated antigens [4]

Serum antibody response to SMP30 in various patients using the methods of Western-blot and ELISA and showed that antibody to SMP30 existed mainly in HCC patients (39.8%), especially in the one with alpha-fetoprotein (AFP) negative

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed cases of HCC (be based on NCCN guidelines triphasic CT and AFP or liver biopsy)
2. Adult patients
3. Both genders are eligible.
4. Informed consent obtained from subject or subject's legal representative

Exclusion Criteria:

1. Patient with other malignancies.
2. Patients with advanced comorbidities except for renal failure.
3. Prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients will be subjected to the following:
  * Detailed History taking.
  * Physical examination.
  * Routine laboratory investigations essential for diagnosis and follow up of patients including:
    1. Complete blood count (CBC).
    2. Chemistry profile: serum bilirubin-serum albumin-SGPT-SGOT.
    3. serum regucalcin(SMP30) antibodies using ELISA
    4. AFP level.
  * Radiological assessment:
  US, Triphasic CT to assess (tumor site, size, numbers, nodal metastases, distal metastases, portal vein invasion..)
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
serum regucalcin in HCC patients | 1-12-2016 to 1-12-2017
  This work aims to assess serum regucalcin antibodies level using ELISA in HCC patients to:
  * evaluate its potential role as biomarker in diagnosis.
  * evaluate potential associations of the presence of serum regucalcin antibody with HCC patients' clinico-epidemiological parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Center Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://ocmu.mans.edu.eg/en/